CLINICAL TRIAL: NCT02126865
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Doses of BI 1060469 Tablets in Healthy Subjects and Otherwise Healthy Patients With Asthma up to GINA Treatment Step 2 (Phase I, Randomised, Placebo-controlled, Double-blind Within Dose Groups)
Brief Title: Multiple Rising Oral Doses of BI 1060469 in Healthy Subjects and Mild Asthma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1333.2; 2013-005463-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (4):
- BI 1060469 Healthy (Experimental): Multiple rising dose qd for 15 days
  Interventions: Drug: BI 1060469 Healthy
- Placebo to BI 1060469 (Placebo Comparator): Matching placebo as tablet for 15 days
  Interventions: Drug: Placebo to BI 1060469
- BI 1060469 asthmatics (Experimental): Multiple rising dose qd for 29 days
  Interventions: Drug: BI 1060469 asthmatics
- Placebo to BI 1060469 asthmatics (Placebo Comparator): Matching placebo as tablet for 29 days
  Interventions: Drug: Placebo to BI 1060469 asthmatics

INTERVENTIONS:
Drug: Placebo to BI 1060469 — tablet
  Arms: Placebo to BI 1060469
Drug: BI 1060469 Healthy — tablet
  Arms: BI 1060469 Healthy
Drug: Placebo to BI 1060469 asthmatics — tablet
  Arms: Placebo to BI 1060469 asthmatics
Drug: BI 1060469 asthmatics — tablet
  Arms: BI 1060469 asthmatics

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1060469 in healthy male and female subjects after oral administration of repeated rising doses of 3 mg, 10 mg, 25 mg, 75 mg, 150 mg and 250 mg qd. of 1 day followed by 14 days and in asthmatic male and female patients after oral administration of repeated rising doses of 25 mg and 150 mg qd of 1 day followed by 28 days.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality, dose linearity after single and multiple dose segments, pharmacodynamics (PD) of BI 1060469 and to describe the PK/PD relationship.

ELIGIBILITY:
Inclusion criteria:

1. Healthy or otherwise healthy asthmatic male or female subjects according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination,vital signs (BP, PR),12-lead ECG, and clinical laboratory tests

   Amended part under fed conditions:

   Healthy female subjects according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (BP, PR),12-lead ECG, and clinical laboratory tests.
2. Age 18 to 55 years (incl.)
3. BMI 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
5. Male subjects,or females who meet any of the following criteria from at least 30 days before the first study drug administration and until 30 days after trial completion:

   * surgically sterilised (including hysterectomy)
   * postmenopausal defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

   Amended part under fed conditions:

   Female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:
   * Use of adequate contraception, e.g. any of the following methods plus condom: implants,injectables,combined oral or vaginal contraceptives,intrauterine device
   * Sexually abstinent
   * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
   * Surgically sterilised (including hysterectomy)
   * Postmenopausal,defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory) In addition for otherwise healthy asthmatic patients
6. Females (of non-child bearing potential) & males,who have a diagnosis of asthma by a physician at least 3 months prior to screening.The diagnosis of asthma must be according to the 2010 Global Initiative for Asthma (GINA) guidelines
7. Pre-bronchodilator clinic measured FEV1 =70% of predicted normal (calculated according to NHANES) measured =6 hours after the last use of short acting bronchodilator at Visit 1 or on the day of randomisation
8. Improvement in FEV1 =12% above baseline or an absolute change of at least 200ml within 15-30 minutes after administration of 400 µg salbutamol. Reversibility testing may be repeated twice during the screening period.At minimum reversibility must have been documented within 12 months prior to inclusion.In case airway reversibility cannot be demonstrated subjects may be entered on the basis of a documented valid mannitol challenge test or proven methacholine- or histamine induced airway hyperreactivity according to ATS,which has to be demonstrated within the last 12 months prior to randomisation
9. Diagnosis of asthma must have been made before the subject's age of 40.If the subject is =40 years and the diagnosis has not yet been recorded in the subject's medical files, the investigator should assess whether the subject's medical history (e.g. symptoms and prescribed medications) confirms the subject suffered from asthma since before the age of 40.If so,this subject may be considered for inclusion after consultation with the Clinical Monitor Local (CML)
10. Subject must have stable asthma not exceeding 8 puffs of salbutamol/day on two consecutive days or 12 puffs/ day between inclusion and randomisation

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator other than asthma up to GINA treatment step 2 or atopic diseases
2. Repeated measurement of systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, or pulse rate outside the range of 50 to 90 mmHg
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Serum creatinine laboratory value out of the normal range
5. GFR according to CKD-EPI-Formula < 80 ml/ min at screening [R12-1392]
6. Current or history of relevant kidney, urinay tract diseases or abnormalities (i.e. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure, infections)
7. Any evidence of a concomitant disease judged clinically relevant by the investigator
8. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
9. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)
10. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders
11. History of relevant orthostatic hypotension, fainting spells, or blackouts
12. Chronic or relevant acute infections
13. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
14. Intake of drugs with a long half-life (greater than 24 hours) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
15. Intake of any NSAIDs, COX2 inhibitors, aspirin, ACE-inhibitors, H2- blockers or OTCor nutripharmaceuticals between screening examination and drug administration
16. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
17. Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication
18. Persons who are committed to an institution by way of official or juridical order will not be enrolled in the study.
19. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
20. Inability to refrain from smoking on specified trial days
21. Alcohol abuse (consumption of more than 20 g/day in females and 30 g/day in males)
22. Drug abuse or positive drug screen
23. Blood donation (more than 100 mL within 30 days prior to administration of trial medication or intended during the trial)
24. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
25. Inability to comply with dietary regimen of trial site
26. At screening, a marked baseline prolongation of QT/QTc interval (such as repeated demonstration of a QTc interval greater than 450 ms) or any other relevant ECG finding
27. A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
28. Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

    For female subjects:

    Exclusion criterion 29 not applicable for the amended part of the study
29. Females who are not surgically sterilised or are not postmenopausal defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)
30. Positive pregnancy test
31. Lactation

    In addition for otherwise healthy asthmatic patients:
32. Any evidence of a clinically relevant concomitant disease other than asthma or atopic diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of subjects with drug-related adverse events (AEs) | Day 1 to 29 or Day 1 to Day 43 (end of trial)

SECONDARY OUTCOMES:
AUCt,1 (area under the concentration-time curve of BI 1060469 in plasma over a uniform dosing interval t after administration of the first dose) | 0 to 672 hours or 0 to 1008 hours
AUC0-infinity (area under the concentration-time curve of BI 1060469 in plasma over the time interval from 0 extrapolated to infinity) | 0 to 672 hours or 0 to 1008 hours
Cmax (maximum measured concentration of BI 1060469 in plasma) | 0 to 672 hours or 0 to 1008 hours
AUCt,ss (area under the concentration-time curve of BI 1060469 in plasma at steady state over a uniform dosing interval t) | 0 to 672 hours or 0 to 1008 hours
Cpre,N (predose concentration of BI 1060469 in plasma immediately before administration of the Nth dose after N-1 doses were administered) | 0 to 672 hours or 0 to 1008 hours
Cmax,ss (maximum measured concentration of BI 1060469 in plasma at steady state) | 0 to 672 hours or 0 to 1008 hours
Linearity index (LI) | 0 to 672 hours or 0 to 1008 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1333.2.1 Boehringer Ingelheim Investigational Site, Berlin, Germany